CLINICAL TRIAL: NCT00764036
Title: Prospective Open Uncontrolled Phase I Study of Compatibility, Safety&Pharmacokinetics of Artesunate, a Semisynthetic Derivative of Artemisinin From the Chinese Herb Artemisia Annua in Patients With Metastatic/Locally Advanced Breast Cancer
Brief Title: Study of Artesunate in Metastatic Breast Cancer
Acronym: ARTIC-M33/2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Hector-Stiftung (Other); Dafra Pharma (Industry); Monika-Kutzner Stiftung, Berlin, Germany (Unknown); HEIFAN-Heidelberger Förderverein d. Ambulanz f. Naturheilkunde eV, Heidelberg, Germany (Unknown)
Responsible Party: Principal Investigator, Cornelia von Hagens, Head Complementary & Integrative Medicine, Dep. 4.2, Heidelberg University
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M33/2
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Breast Cancer; Locally Advanced Breast Cancer
Keywords: phase I; safety
MeSH Terms: conditions — Breast Neoplasms | interventions — Artesunate

STUDY DESIGN:
Intervention Model Description: dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm only (Experimental): add-on therapy with 100, 150 or 200 mg oral artesunate once daily
  Interventions: Drug: artesunate

INTERVENTIONS:
Drug: artesunate — add-on therapy with daily single oral doses of 100, 150 or 200 mg of artesunate
  Other Names: artesunic acid hemisuccinate; dihydroqinghaosu hemisuccinate

SUMMARY:
The purpose of this study is to evaluation the tolerability of an add-on therapy with artesunate with a duration of 4 weeks in patients with advanced breast cancer.

DETAILED DESCRIPTION:
Additional objectives are:

* parallel sampling of blood and saliva for the determination of drug concentrations and pharmacokinetic parameters in a substudy on the day of first application and during steady state
* attempt to establish a therapeutical drug monitoring
* collection of further safety data during prolonged add-on treatments (compassionate use)

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed breast cancer
* Distant metastases or locally advanced breast cancer
* Age ≥ 18 years
* ECOG performance ≤ 2
* Life expectancy of at least 6 months
* Written informed consent
* individual standard therapy according to guidelines
* Oral intake of trial medication possible
* Compliance with study procedures
* Women of childbearing potential: negative pregnancy test before start of medication
* Use of a highly effective method of birth control during intake of add-on therapy for women of childbearing potential being sexually active

Inclusion Criteria for Extended Treatment Phase:

* Participant of the phase I study ARTIC M33/2 who had tolerated the study medication for 4±1 weeks without clinically relvant adverse events or after improvement to ≤ grade 2
* Participant of the phase I study ARTIC M33/2 with possible benefit by continuation or restart of the add-on therapy after a next progression according to current scientific knowledge
* Written informed consent for extended treatment phase
* Consent of the responsible oncologist
* Compliance for further intake and follow-up expected

Inclusion Criteria for Individual Compassionate Use:

* Participant of the phase I study ARTIC M33/2
* Available standard therapies have minimal or only short activity or intolerable side effects
* Written informed consent for compassionate use
* Consent of the responsible oncologist

Exclusion Criteria:

* Allergy to artesunate or to other artemisinin derivatives
* Concurrent conditions interfering with patient safety
* Communication problems
* Concurrent participation in another clinical trial or 4 weeks prior to recruitment
* Participation in a clinical trial with an unapproved drug 6 months prior to recruitment
* Sinus bradycardia, bradyarrhythmia
* AV-Block II° and III°
* QTc > 500 msec
* Previously known long QT-syndrome
* Concurrent intake of a medication with clinically relevant neurotoxicity or during 30 days prior to recruitment
* Relevant neurological symptoms which might complicate the evaluation of the compatibility of the IMPD (f. e. cerebral metastases) or might be subject to worsening during intake of the IMPD
* Radiotherapy 2 weeks prior of the intake of the IMPD
* Concurrent intake of supplements or any other medication with unapproved efficacy f.e. vitamins, minerals or others (OTC)
* Pregnancy and lactation
* Ineffective mode of contraception in women of childbearing potential

Exclusion Criteria for Extended Treatment Phase:

* Clinically relevant adverse Events during the first 4 weeks of intake of study medication possibly, probably or definitely related to the study medication
* Intolerable health risks by continuation re-exposition with the study medication
* Continuation or re-exposition is medically not acceptable after consultation of physicians responsible for their standard therapy

Exclusion Criteria for Individual Compassionate Use:

- Intolerable health risks by re-exposition with the study medication

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Dose limiting adverse events with possible, probable or definite relation with the respective dose level of the add-on therapy | 8-12 weeks

SECONDARY OUTCOMES:
Adverse events relation between adverse events and add-on therapy, cortisol profile in saliva, overall response rate, clinical benefit, assessment of patients expectations | 8-12 weeks

OTHER OUTCOMES:
Further safety data (adverse events) during prolonged treatments latest till the second progression during the add-on therapy with the study medication (compassionate use) | add-on treatments > 4+/- 1 weeks
Collection of further safety data during later individual compassionate use with monitoring if approbriate for the patients' health status | Depending on patients' preference and health status

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia U v. Hagens, MD, Principal Investigator — Department of Gynecological Endocrinology and Reproductive Medicine
Locations (1):
- Complementary and Integrative Medicine, Dep. Gyn. Endocrinology, Women's Hospital, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birgersson S, Ericsson T, Blank A, Hagens Cv, Ashton M, Hoffmann KJ. A high-throughput LC-MS/MS assay for quantification of artesunate and its metabolite dihydroartemisinin in human plasma and saliva. Bioanalysis. 2014 Sep;6(18):2357-69. doi: 10.4155/bio.14.116. PMID 25384589
- [Result] von Hagens C, Walter-Sack I, Goeckenjan M, Osburg J, Storch-Hagenlocher B, Sertel S, Elsasser M, Remppis BA, Edler L, Munzinger J, Efferth T, Schneeweiss A, Strowitzki T. Prospective open uncontrolled phase I study to define a well-tolerated dose of oral artesunate as add-on therapy in patients with metastatic breast cancer (ARTIC M33/2). Breast Cancer Res Treat. 2017 Jul;164(2):359-369. doi: 10.1007/s10549-017-4261-1. Epub 2017 Apr 24. PMID 28439738
- [Result] Konig M, von Hagens C, Hoth S, Baumann I, Walter-Sack I, Edler L, Sertel S. Investigation of ototoxicity of artesunate as add-on therapy in patients with metastatic or locally advanced breast cancer: new audiological results from a prospective, open, uncontrolled, monocentric phase I study. Cancer Chemother Pharmacol. 2016 Feb;77(2):413-27. doi: 10.1007/s00280-016-2960-7. Epub 2016 Jan 21. PMID 26793976
- [Result] Konig M, von Hagens C, Hoth S, Baumann I, Walter-Sack I, Edler L, Sertel S. Erratum to: Investigation of ototoxicity of artesunate as add-on therapy in patients with metastatic or locally advanced breast cancer: new audiological results from a prospective, open, uncontrolled, monocentric phase I study. Cancer Chemother Pharmacol. 2016 Jun;77(6):1321. doi: 10.1007/s00280-016-3023-9. No abstract available. PMID 27094900
- [Result] Ericsson T, Blank A, von Hagens C, Ashton M, Abelo A. Population pharmacokinetics of artesunate and dihydroartemisinin during long-term oral administration of artesunate to patients with metastatic breast cancer. Eur J Clin Pharmacol. 2014 Dec;70(12):1453-63. doi: 10.1007/s00228-014-1754-2. Epub 2014 Sep 25. PMID 25248945